CLINICAL TRIAL: NCT00679406
Title: Treatment of Insomnia in Military Veterans:Phase 1
Brief Title: Brief Behavioral Treatment of Insomnia in Military Veterans: Phase 1
Acronym: BBTIMV1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anne Germain, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO07110063; NIMH: 1 R34 MH080696
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Insomnia
Keywords: Chronic Insomnia lasting more than 1 month
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Brief Behavioral Treatment for Insomnia
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia — Effective behavioral insomnia treatments are typically delivered over an 8-week period. This format may not be easily exportable to primary and community care settings where military returnees and veterans seek help. The goal here is to test the effects of a 4-week behavioral treatment that targets chronic insomnia (lasting >1 month) in service members returning from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF), and who present with the typical psychiatric comorbidities associated of combat-related anxiety and mood disorders and stress reactions.
  Other Names: BBTI

SUMMARY:
The purpose of this study is to adapt and test the effects of a 4-week behavioral treatment that targets chronic insomnia (lasting >1 month) in service members returning from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF).

DETAILED DESCRIPTION:
Insomnia is one of the most common reasons for referral to mental health services in active duty personnel. Chronic insomnia often persists post-deployment, contributes to poor mental and physical health outcomes, and requires targeted interventions. Effective behavioral treatments of insomnia have not been adapted and tested for the treatment of chronic insomnia comorbid to combat-related mental disorders and stress reactions. In addition, effective behavioral insomnia treatments are typically delivered over an 8-week period. This format may not be easily exportable to primary and community care settings where military returnees and veterans seek help. The goal of this R34 Exploratory Clinical Research Grant is to adapt and test the effects of a 4-week behavioral treatment that targets chronic insomnia (lasting >1 month) in service members returning from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF), and who present with the typical psychiatric comorbidities associated of combat-related anxiety and mood disorders and stress reactions. We call this intervention the Brief Behavioral Treatment of Insomnia for Military Veterans (BBTI-MV). The proposed study includes two phases. Phase I aims at iteratively adapting and refining a treatment manual for insomnia in OIF/OEF military returnees. Outcomes of interest include self-report, diary, and actigraphic sleep measures, as well as measures of PTSD, anxiety, and depression, and perceived physical health.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18 and older.
2. Military returnees from OIF/OEF
3. Meet diagnostic criteria for chronic insomnia as defined by:

   * a. Complaint of sleep latency >30 minutes, or wake time after sleep onset >30 minutes, or Sleep Efficiency <85%, or a complaint of non-restorative sleep;
   * b. Frequency of insomnia complaint >3 times per week;
   * c. Duration of insomnia complaint >1 month
   * d. Associated with at least one daytime consequences
4. If using sleep medications, medication and dosage have not been changed in the past month, and will remain unchanged for the duration of the acute treatment phase of the study (i.e., 4 weeks)
5. If using other psychotropic medications, medication and dosage have not been changed in the past 2 months, and will remain unchanged for the duration of the acute treatment phase of the study (i.e., 4 weeks)

Exclusion Criteria:

1. Active duty personnel, or reservists/national guards scheduled for re-deployment over the following eight months
2. Untreated, current, and severe PTSD as determined on the SCID.
3. Untreated, current, and severe Major Depressive Disorder as determined by the Structured Clinical Interview for DSM-IV and a score > 30 on the Beck Depression Inventory
4. Psychotic or bipolar disorder
5. Current substance or alcohol use disorder as determined by the SCID or by positive drug toxicology results
6. Unstable medical condition
7. Hospitalization in the previous 2 weeks for a medical condition or surgery for which recovery overlaps with the study onset and duration
8. Seizure disorder or traumatic brain injury.
9. Current sleep disorders such as nightmare disorder, restless legs syndrome, or suspected sleep disorder requiring polysomnographic assessment, such as obstructive sleep apnea or periodic leg movements.
10. Sleep apnea revealed during the screening sleep study.
11. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Diary | Weekly during entire participation
Pittsburgh Sleep Quality Index (PSQI) | Baseline and Post Intervention
PSQI Addendum for PTSD (PSQIA) | Baseline and Post Intervention
Sleep quality defined by:PIRS 20 and the ISI | Screening, Baseline, and Post Intervention

SECONDARY OUTCOMES:
PTSD symptom severity as measured by the CAPS | Screening
Depression: BDI | Baseline and Post Intervention
Anxiety: BAI | Baseline and Post Intervention
Medical History: MHQ, MEDHIST_2WK, MOS | Screening, Baseline, and Post Intervention
Trauma History: THQ,CES,PCL-C,ICG | Screening, Baseline, and Post Intervention
Post Sleep Self Report: PSEQ-SV and POST | Screening
Sleepiness: EPWORTH, BASS | Screening, Baseline, and Post Intervention
Expectations and Satisfaction: TEQ-94, Client Satisfaction Survey | Baseline and Post Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anne Germain, PhD., Principal Investigator — University of Pittsburgh, Department of Psychiatry
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States